CLINICAL TRIAL: NCT06573606
Title: Ophthalmic Solution in Diabetic Corneal Alteration
Status: Completed | Type: Observational
Sponsor: D&V FARMA srl (Industry)
Collaborators: San Giovanni Addolorata Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DIDI01
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HA-CS: Diabetic subjects affected by dry eye disease are treated with the new ophthalmic solution containing cross-linked hyaluronic acid (CX-HA) and Chondroitin sulphate (CS).
  Interventions: Device: CX-HA and CS

INTERVENTIONS:
Device: CX-HA and CS — Sterile Isotonic ophthalmic solution

SUMMARY:
Data analyses and revision of the DED symptoms in diabetic subjects. A novel ophthalmic solution containing cross-linked ha (CX-HA) and Chondroitin sulphate (CS) has been made available on the market.

Both molecules have been widely studied for their viscoelastic and hydrating properties.

Nevertheless, the use of CS in ophthalmology has been limited since, routinely, the molecule is of animal origins.

This new ophthalmic solution is the first on the market formulated with a CS of non-animal origin.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Subjects affected by dry eye disease

Exclusion Criteria:

* know allergies to CX-HA
* know allergies to CS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data derived from diabetic subject affected by dry eye disease and treated with the ophthalmic solution containing CX-HA and CS will be collected and analysed
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
TBUT | 3 months
  Tear Breakup Time

SECONDARY OUTCOMES:
OSDI | 3 months
  Ocular Surface Disease Index
Corneal Sensitivity | 3 months
  measured via the "Luneau Cochet-Bonnet Aesthesiometer", results are expressed in cm
Wound Healing | 30 hours
  Scratch test performed on cell lines using the "Ibidi Culture-Inserts". The test provides hinds on the ability of a cell line to cover a "wound" created in the monolayer. Results are given as % of the area covered

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni-Addolorata Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zou X, Lu L, Xu Y, Zhu J, He J, Zhang B, Zou H. Prevalence and clinical characteristics of dry eye disease in community-based type 2 diabetic patients: the Beixinjing eye study. BMC Ophthalmol. 2018 May 10;18(1):117. doi: 10.1186/s12886-018-0781-7. PMID 29747621
- [Background] Guerrero-Moreno A, Baudouin C, Melik Parsadaniantz S, Reaux-Le Goazigo A. Morphological and Functional Changes of Corneal Nerves and Their Contribution to Peripheral and Central Sensory Abnormalities. Front Cell Neurosci. 2020 Dec 10;14:610342. doi: 10.3389/fncel.2020.610342. eCollection 2020. PMID 33362474
- [Background] Yoo TK, Oh E. Diabetes mellitus is associated with dry eye syndrome: a meta-analysis. Int Ophthalmol. 2019 Nov;39(11):2611-2620. doi: 10.1007/s10792-019-01110-y. Epub 2019 May 7. PMID 31065905
- [Background] Posarelli C, Passani A, Del Re M, Fogli S, Toro MD, Ferreras A, Figus M. Cross-Linked Hyaluronic Acid as Tear Film Substitute. J Ocul Pharmacol Ther. 2019 Sep;35(7):381-387. doi: 10.1089/jop.2018.0151. Epub 2019 Aug 2. PMID 31373862
- [Background] Ledbetter EC, Munger RJ, Ring RD, Scarlett JM. Efficacy of two chondroitin sulfate ophthalmic solutions in the therapy of spontaneous chronic corneal epithelial defects and ulcerative keratitis associated with bullous keratopathy in dogs. Vet Ophthalmol. 2006 Mar-Apr;9(2):77-87. doi: 10.1111/j.1463-5224.2006.00439.x. PMID 16497231
- [Background] Postorino EI, Rania L, Aragona E, Mannucci C, Alibrandi A, Calapai G, Puzzolo D, Aragona P. Efficacy of eyedrops containing cross-linked hyaluronic acid and coenzyme Q10 in treating patients with mild to moderate dry eye. Eur J Ophthalmol. 2018 Jan;28(1):25-31. doi: 10.5301/ejo.5001011. Epub 2018 Feb 19. PMID 28777385
- [Background] Carlson E, Kao WWY, Ogundele A. Impact of Hyaluronic Acid-Containing Artificial Tear Products on Reepithelialization in an In Vivo Corneal Wound Model. J Ocul Pharmacol Ther. 2018 May;34(4):360-364. doi: 10.1089/jop.2017.0080. Epub 2018 Feb 2. PMID 29394128
- [Derived] Scarinci F, De Simone G, Ciancimino C, Caggiano C, Pocobelli G, Di Masi A. Enhancing Corneal Sensitivity in Diabetic Patients Through an Innovative Ophthalmic Solution: In Vivo and Vitro Results. J Clin Med. 2025 Jan 3;14(1):245. doi: 10.3390/jcm14010245. PMID 39797325